CLINICAL TRIAL: NCT06015932
Title: A Non-Randomized Translational Trial of Cognitive Behavioral Cancer Stress Management (CBCSM) and Its Effects on Cancer Distress
Brief Title: Group Cognitive Behavior Sessions (CBCSM) to Decrease Distress in Cancer Patients
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Shawna L. Ehlers, Ph.D., L.P., Principal Investigator, Mayo Clinic
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 17-000947; NCI-2023-00250 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 17-000947 (Other: Mayo Clinic)
Record Dates: First submitted 2023-08-23; First posted 2023-08-29 (Actual); Last update posted 2025-07-29 (Actual); Status verified 2025-07

CONDITIONS: Hematopoietic and Lymphoid System Neoplasm; Malignant Solid Neoplasm; Metastatic Malignant Solid Neoplasm
MeSH Terms: conditions — Neoplasm Metastasis | interventions — Cognitive Behavioral Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Group I (CBCSM) (Experimental): Patients participate in five CBCSM group sessions on study. Patients complete questionnaires throughout the trial and during follow-up at 1, 3, 6, and 12 months.
  Interventions: Behavioral: Cognitive Behavior Therapy; Other: Questionnaire Administration
- Group II (no CBCSM) (Active Comparator): Patients complete questionnaires throughout the trial and during follow-up at 1, 3, 6, and 12 months.
  Interventions: Other: Questionnaire Administration

INTERVENTIONS:
Behavioral: Cognitive Behavior Therapy — Participate in CBCSM group sessions
  Other Names: CBT; cognitive therapy; CT
  Arms: Group I (CBCSM)
Other: Questionnaire Administration — Complete questionnaires

SUMMARY:
This clinical trial tests how well cognitive behavioral cancer stress management (CBCSM) group sessions work to decrease psychological distress in cancer patients. CBCSM teaches patients how to recognize and reduce the impacts of cancer associated stress on the biological, psychological, and social life domains.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To reduce psychological stress.

SECONDARY OBJECTIVES:

I. To increase post-traumatic growth (PTG). II. To increase patient self-efficacy in utilizing therapy skills. III. To estimate patient acceptability and feasibility of conducting CBCSM within the clinical setting.

IV. To estimate differences of conducting CBCSM virtually during the Public Health Emergency (PHE) versus in person pre-PHE.

V. To estimate differences of conducting CBCSM post PHE virtually with limitation to Minnesota patients only.

VI. To explore the difference using the same therapy in patients with advanced, metastatic disease in a individual setting versus patients without the advanced, metastatic disease in a group setting.

OUTLINE: Patients are assigned to 1 of 2 groups.

GROUP I: Patients participate in five CBCSM group sessions on study. Patients complete questionnaires throughout the trial and during follow-up at 1, 3, 6, and 12 months.

GROUP II: Patients complete questionnaires throughout the trial and during follow-up at 1, 3, 6, and 12 months.

ELIGIBILITY:
Inclusion Criteria:

* Eligible for the cognitive behavioral cancer stress management (CBCSM) clinical service
* Cancer diagnosis with predicted survival > 1 year
* Cancer treatment within past 1 year or treatment planning in progress
* Age >= 18-years
* Moderate distress screen, indicated by Impact of Event Scale-Revised (IES-R) score >= 14 or clinical judgment
* Written informed research consent

Exclusion Criteria:

* Inability to actively participate in and learn from group therapy (e.g., psychotic symptoms, neurological condition, personality pathology) as determined by clinical judgment in clinical consultation (Individual therapy or alternative group therapy will be offered)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 400 (Estimated)
Dates: Start 2017-12-20 (Actual); Primary Completion 2029-12 (Estimated); Study Completion 2029-12 (Estimated)

PRIMARY OUTCOMES:
Change in post-traumatic stress (PTS) score | At baseline, 1, 3, 6, and 12 months
  Each item on the PTS is rated on a 5-point scale (0=Not at all; 1=A little bit; 2=Moderately; 3=Quite a bit, and 4=Extremely). The total score can range from 0 to 36 with higher scores indicating greater severity of posttraumatic stress disorder.

SECONDARY OUTCOMES:
Change in post-traumatic growth (PTG) score | At baseline, 1, 3, 6, and 12 months
  PTG will be assessed using the Patient-Reported Outcomes Measurement System (PROMIS®)-Psychosocial Impact Scale-Positive. The PROMIS assesses pain intensity using a single 0-10 numeric rating item and seven health domains (physical function, fatigue, pain interference, depressive symptoms, anxiety, ability to participate in social roles and activities, and sleep disturbance) using four items per domain.
Change in self-efficacy score | At baseline, 1, 3, 6, and 12 months
  Will examine predicted increase in self-efficacy associated with Cognitive Behavioral Cancer Stress Management (CBCSM) from pre-intervention to post-intervention. Scores will be assessed using the Measure of Current Status-Part A (MOCS-A), which measures participants' current self-perceived status on several skills: the ability to relax at will, recognize stress-inducing situations, restructure maladaptive thoughts, be assertive about needs, express anger effectively and appropriately, and choose appropriate coping responses as needed. Ratings are made on a scale from I cannot do this at all (0) to I can do this extremely well (4).
Patient acceptability and satisfaction | Baseline to 12 months
  Will be assessed by simple percentage, based on scores from an Institute for Healthcare Improvement 10-point Likert scale (0-10, "Would you recommend this program to your friends and family?" A score ≥7 indicates high individual satisfaction.
Patient attendance and feasibility | Baseline to 12 months
  Will be assessed by simple percentage. Attendance and feasibility will be determined by the number of patients attending ≥3 sessions out of five.
Anxiety | At baseline, 1, 3, 6, and 12 months
  Will examine predicted reductions in anxiety symptoms associated with Cognitive Behavioral Cancer Stress Management (CBCSM) from pre-intervention to post-intervention. Anxiety will be measured using General Anxiety Disorder-7 (GAD-7) symptom scores, an 8-question survey. Seven questions are answered on a 0-3 scale where 0=Not at all and 3=Nearly every day. The final question is answered on a 4-point scale from Not Difficult at All to Extremely Difficult.
Depression | At baseline, 1, 3, 6, and 12 months
  Will examine predicted reductions in depression symptoms associated with Cognitive Behavioral Cancer Stress Management (CBCSM) from pre-intervention to post-intervention. Level of depression will be determined using the Patient Health Questionnaire-8 (PHQ-8). The PHQ-8 is an 8-item questionnaire answered on a scale of 0-3 where 0=Not at all and 3=Nearly every day.

CONTACTS AND LOCATIONS:
Overall Officials: Shawna L. Ehlers, Ph.D., L.P., Principal Investigator — Mayo Clinic in Rochester
Locations (1):
- Mayo Clinic in Rochester, Rochester, Minnesota, United States

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials